CLINICAL TRIAL: NCT01103687
Title: A Phase 1 Randomized, Double-Blind, Placebo Controlled Clinical Trial to Evaluate the Safety, Mucosal Immunogenicity and Innate Immune Responses of Recombinant Adenovirus Serotype 26 HIV-1 Vaccine (Ad26.ENVA.01) in Healthy, HIV-1 Uninfected Adults (Ad26.ENVA.01 (rAd26) HIV-1 Mucosal/IPCAVD-003 Vaccine Study)
Brief Title: Evaluating the Safety and Immune Response of an Adenovirus-Based HIV Vaccine in HIV-Uninfected Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Ad26.ENVA.01 Mucosal/IPCAVD003; 11678 (Registry Identifier: DAIDS ES Registry ID); Ad26.ENVA.01 Mucosal; Ad26.ENVA.01Mucosal/IPCAVD-003
Record Dates: First submitted 2010-04-13; First posted 2010-04-15 (Estimated); Last update posted 2017-09-08 (Actual); Status verified 2017-09

CONDITIONS: HIV Infections
Keywords: HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ad26.ENVA.01 (rAd26) (Experimental): Participants will receive the Ad26.ENVA.01 (rAd26) vaccine at baseline.
  Interventions: Biological: Ad26.ENVA.01 (rAd26)
- Placebo Vaccine (Placebo Comparator): Participants will receive the placebo vaccine at baseline.
  Interventions: Biological: Placebo Vaccine

INTERVENTIONS:
Biological: Ad26.ENVA.01 (rAd26) — 5 x 10^10 virus particles (VP) vaccine delivered intramuscularly (IM)
  Arms: Ad26.ENVA.01 (rAd26)
Biological: Placebo Vaccine — Placebo vaccine delivered IM
  Other Names: FFB, final formula buffer
  Arms: Placebo Vaccine

SUMMARY:
The purpose of this study is to evaluate the safety and immune response of an adenovirus-based HIV vaccine in HIV-uninfected adults.

DETAILED DESCRIPTION:
Control of the global HIV pandemic will require the development of a safe and effective vaccine. Many HIV preventive vaccines that are in development use a recombinant adenovirus serotype 5 (rAd5) vector as a way of delivering the vaccine into cells. However, the majority of people, particularly in the developing world, have immunity against the Ad5 vector, which means the vaccine will not be effective at preventing HIV infection. This study will use a rAd26 vector as part of a HIV vaccine, as research has shown that relatively few people have immunity against this vector. The purpose of this study is to evaluate the safety and immunogenicity of a rAd26 vector preventive HIV-1 vaccine.

This study will enroll healthy, HIV-uninfected people. Participants will be randomly assigned to receive either the rAd26 vaccine or a placebo vaccine. All vaccines will be injected into the upper arm. At the vaccination study visit, participants will undergo a medical and medication history review, physical examination, and a rectal sampling procedure. They will then receive their assigned vaccine. After receiving the vaccine, participants will remain in the clinic for at least 30 minutes for observation and monitoring of side effects. Participants will receive counseling on HIV risk reduction and pregnancy prevention. For 7 days after the vaccination, participants will monitor their temperature and side effects. Additional study visits will occur at Days 1, 3, 7, 14, 28, 61, 168, and 365. At these visits, participants will undergo a medical history review, physical examination, counseling, and blood collection. At the Day 14 and 168 visits, a rectal sampling procedure will be performed. Participants will attend a study visit or be contacted by study researchers by telephone or e-mail 18 months after receiving the vaccine for follow-up health and safety monitoring. Participants may elect to attend optional follow-up visits for blood collection at Years 2, 3, 4, and 5.

ELIGIBILITY:
Inclusion Criteria:

* Willing to be followed for the planned duration of the study
* Able and willing to provide informed consent
* Assessment of understanding, including the completion of a questionnaire prior to vaccination; verbally demonstrated understanding of all questionnaire items answered incorrectly
* Willing to receive HIV test results
* In good general health as shown by medical history, physical exam, and screening laboratory tests
* Hemoglobin levels greater than or equal to 11.0 g/dL for women and greater than or equal to 12.5 g/dL for men
* White blood cell (WBC) count between 3,300 and 12,000 cells/mm3
* Total lymphocyte count greater than or equal to 800 cells/mm3
* Remaining differential either within institutional normal range or accompanied by site physician approval
* Platelet levels between 125,000 and 550,000/mm3
* Alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase, and total bilirubin less than 1.25 times the institutional upper limit of normal; and creatinine less than or equal to the institutional upper limit of normal
* Negative HIV-1 and 2 blood test
* Negative hepatitis B surface antigen (HBsAg)
* Negative anti-hepatitis C virus antibodies (anti-HCV), or negative HCV polymerase chain reaction (PCR) if the anti-HCV is positive
* Normal urine test; more information about this criterion can be found in the protocol
* Female participants must have a negative serum or urine beta human chorionic gonadotropin (β-HCG) pregnancy test performed on the day of vaccination prior to vaccination
* Female participants must agree to consistently use contraception from at least 21 days prior to study entry through the last study visit. More information on this criterion can be found in the protocol.

Exclusion Criteria:

* Received HIV vaccine(s) in a prior HIV vaccine trial. Participants who received a control/placebo in an HIV vaccine trial are not excluded but documentation of the identity of the study control/placebo must be obtained.
* Immunosuppressive medications received within 168 days before vaccination (e.g., oral/parenteral corticosteroids, and/or cytotoxic medications). People taking corticosteroid nasal spray for allergic rhinitis and topical corticosteroids for mild, uncomplicated dermatitis are not excluded.
* Blood products received within 120 days before vaccination
* Immunoglobulin received within 60 days before vaccination
* Live attenuated vaccines received within 30 days before vaccination (e.g., measles, mumps, and rubella [MMR]; oral polio vaccine [OPV]; varicella; yellow fever; Flumist® influenza)
* Investigational research agents received within 30 days before vaccination
* Any vaccines that are not live attenuated vaccines and were received within 14 days prior to vaccination (e.g., influenza, tetanus, pneumococcal, Hepatitis A or B)
* Clinically significant medical condition, physical examination findings, clinically significant abnormal laboratory results, or past medical history with clinically significant implications for current health. More information on this criterion can be found in the protocol.
* Any medical, psychiatric, or social condition, or occupational or other responsibility that, in the judgment of the investigator, would interfere with, or serve as a contraindication to, protocol adherence, assessment of safety or reactogenicity, or a participant's ability to give informed consent
* Serious adverse reactions to vaccines including anaphylaxis and related symptoms such as hives, respiratory difficulty, angioedema, and/or abdominal pain. People who had a nonanaphylactic adverse reaction to the pertussis vaccine as a child are not excluded.
* Known autoimmune disease
* Known immunodeficiency
* Active syphilis infection. People who had syphilis that was fully treated more than 6 months before study entry are not excluded.
* Asthma other than mild, well-controlled asthma. More information on this criterion can be found in the protocol.
* Diabetes mellitus type 1 or type 2, including cases controlled with diet alone. People with a history of isolated gestational diabetes are not excluded.
* Thyroidectomy, or thyroid disease requiring medication in the 12 months before study entry
* Angioedema in the 3 years before study entry if episodes are considered serious or have required medication in the 2 years before study entry
* If a person has been diagnosed with high blood pressure during screening or previously, they will be excluded for high blood pressure that is not well controlled. If a person has NOT been diagnosed with high blood pressure during screening or previously, they will be excluded for systolic blood pressure greater than or equal to 150 mm Hg at study entry or diastolic blood pressure greater than or equal to 100 mm Hg at study entry.
* Body mass index (BMI) greater than or equal to 40, or BMI greater than or equal to 35 and two or more of the following conditions: age greater than 45, systolic blood pressure greater than 140 mm Hg, diastolic blood pressure greater than 90 mm Hg, current smoker, or known hyperlipidemia
* Bleeding disorder diagnosed by a doctor (e.g., factor deficiency, coagulopathy, platelet disorder requiring special precautions)
* Cancer. People with a surgical excision and subsequent observation period that in the investigator's estimation has a reasonable assurance of sustained cure or is unlikely to recur during the study period are not excluded.
* Seizure disorder or experienced a seizure in the 3 years before study entry. People with a history of seizures who have not required medications or had a seizure in the 3 years before study entry are not excluded.
* Absence of a functional spleen
* Psychiatric condition that makes study compliance difficult (e.g., people with psychoses in the 3 years before study entry, ongoing risk for suicide, history of suicide attempt or gesture in the 3 years before study entry)
* Pregnant or breastfeeding
* Abnormality of the rectum or rectal mucosa, which in the opinion of the clinician represents a contraindication to rectal biopsy
* Use of medication interfering with normal coagulation that may increase the risk for bleeding at the time of the rectal biopsy
* Experimental vaccine(s) received in a prior vaccine trial in the 5 years before study entry. Exceptions may be made for vaccines that are currently licensed or have subsequently undergone licensure. For potential participants who have received control/placebo in an experimental vaccine trial, the protocol safety review team (PSRT) will determine eligibility on a case-by-case basis. For potential participants who have received an experimental vaccine(s) more than 5 years ago, eligibility for enrollment will be determined by the PSRT on a case-by-case basis.
* Men who have sex with men (MSM) who have had receptive anal intercourse in the 12 months before study entry must have a positive rectal gonorrhea or chlamydia test by nucleic acid amplification test (NAAT) or culture
* Perianal herpes simplex virus (HSV) outbreak in the 30 days before study entry
* History of newly acquired syphilis, gonorrhea, non-gonococcal urethritis, HSV2, chlamydia, pelvic inflammatory disease (PID), trichomonas, mucopurulent cervicitis, epididymitis, proctitis, lymphogranuloma venereum, chancroid, or hepatitis B in the 12 months prior to study entry
* Individuals who are classified as not low-risk for acquisition of HIV-1 infection, on the basis of sexual behaviors within the 12 months prior to study entry. More information on this criterion can be found in the protocol.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2010-07; Primary Completion 2012-09 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Local and systemic reactions to vaccine | Measured through the 18-month follow-up visit
Adverse and serious adverse experiences | Measured through the 18-month follow-up visit

SECONDARY OUTCOMES:
Innate immune responses, including cytokine levels and natural killer (NK) cell populations | Measured through the 18-month follow-up visit
Humoral immune responses, including neutralizing antibodies against HIV and Ad26 and binding antibodies | Measured through the 18-month follow-up visit
Cell mediated immunity, including T-cell gamma interferon responses by enzyme-linked immunosorbent spot (ELISPOT) and T-cell responses by flow cytometry | Measured through the 18-month follow-up visit
Mucosal immune responses, including histopathology and T-cell responses by flow cytometry | Measured through the 18-month follow-up visit
Genotyping | Measured through the 18-month follow-up visit

CONTACTS AND LOCATIONS:
Overall Officials: Lindsey Baden, Study Chair — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hosp. Novel Adenoviral Vector Prophylactic HIV Vaccine Non-Network CRS, Boston, Massachusetts, United States

REFERENCES:
- [Background] Mast TC, Kierstead L, Gupta SB, Nikas AA, Kallas EG, Novitsky V, Mbewe B, Pitisuttithum P, Schechter M, Vardas E, Wolfe ND, Aste-Amezaga M, Casimiro DR, Coplan P, Straus WL, Shiver JW. International epidemiology of human pre-existing adenovirus (Ad) type-5, type-6, type-26 and type-36 neutralizing antibodies: correlates of high Ad5 titers and implications for potential HIV vaccine trials. Vaccine. 2010 Jan 22;28(4):950-7. doi: 10.1016/j.vaccine.2009.10.145. Epub 2009 Nov 17. PMID 19925902
- [Background] Priddy FH, Brown D, Kublin J, Monahan K, Wright DP, Lalezari J, Santiago S, Marmor M, Lally M, Novak RM, Brown SJ, Kulkarni P, Dubey SA, Kierstead LS, Casimiro DR, Mogg R, DiNubile MJ, Shiver JW, Leavitt RY, Robertson MN, Mehrotra DV, Quirk E; Merck V520-016 Study Group. Safety and immunogenicity of a replication-incompetent adenovirus type 5 HIV-1 clade B gag/pol/nef vaccine in healthy adults. Clin Infect Dis. 2008 Jun 1;46(11):1769-81. doi: 10.1086/587993. PMID 18433307
- [Derived] Baden LR, Liu J, Li H, Johnson JA, Walsh SR, Kleinjan JA, Engelson BA, Peter L, Abbink P, Milner DA Jr, Golden KL, Viani KL, Stachler MD, Chen BJ, Pau MG, Weijtens M, Carey BR, Miller CA, Swann EM, Wolff M, Loblein H, Seaman MS, Dolin R, Barouch DH. Induction of HIV-1-specific mucosal immune responses following intramuscular recombinant adenovirus serotype 26 HIV-1 vaccination of humans. J Infect Dis. 2015 Feb 15;211(4):518-28. doi: 10.1093/infdis/jiu485. Epub 2014 Aug 26. PMID 25165165